CLINICAL TRIAL: NCT05922202
Title: Influence of Frailty on Cardiovascular Events and Mortality in Patients With Chronic Obstructive Pulmonary Disease (COPD): A Multicentre Observational Study.
Brief Title: Influence of Frailty on Cardiovascular Events and Mortality in Patients With COPD.
Acronym: FrCVCOPD
Status: Recruiting | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria di Modena (Other)
Collaborators: Campus Bio-Medico Universitario di Roma-Medicina Interna - Servizio di Pneumologia (Unknown); Ospedale Sant'Andrea - Azienda Sanitaria Locale di Vercelli-Reparto di Pneumologia (Unknown); Hospitals - Aneurin Bevan University Heath Board (Wales) - United Kingdom (Unknown)
Responsible Party: Principal Investigator, Alessia Verduri, Dr Alessia Verduri, Azienda Ospedaliero-Universitaria di Modena
Other Study IDs: 6390
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Role of Frailty in COPD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- COPD outpatients: Outpatients with COPD. COPD diagnosis confirmed by spirometry and according to Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) guidelines.
  Interventions: Other: Assessment of cardiovascular events, cardiovascular mortality, all-cause mortality, and mortality due to COPD at 12 and 24 months

INTERVENTIONS:
Other: Assessment of cardiovascular events, cardiovascular mortality, all-cause mortality, and mortality due to COPD at 12 and 24 months — At 12 and 24 months of follow up, cardiovascular events (including hospital admissions), deaths due to cardiovascular disease, deaths due to all-cause, deaths due to COPD will be recorded in COPD outpatients group.

SUMMARY:
Observational study on the influence of frailty on cardiovascular risk in COPD.

DETAILED DESCRIPTION:
The study will investigate the influence that frailty can have on cardiovascular risk in patients with COPD. The project will assess the association between frailty and all-cause mortality, and the relationship between frailty and cardiovascular mortality, by comparing COPD patients living with frailty vs non-frail COPD patients.

The study participants will be outpatients with diagnosis of COPD according to the Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) guidelines (www.goldcopd.org).

Frailty will be measured using the Clinical Frailty Scale (grades 1-9). Patients who are terminally ill (CFS = 9) will be excluded. Cognitive function will be explored using the Montreal Cognitive Assessment (MoCA) test.

The follow up will be at 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with age ≥18 years, with diagnosis of COPD of at least 1 year, in stable condition, without acute exacerbation in the last 30 days and/or all-cause hospitalisation in the last 3 months
* Smoking history of ≥ 10 pack/years
* Diagnosis of COPD according to GOLD guidelines (www.goldcopd.org)
* Individuals able to provide their written informed consent.

Exclusion Criteria:

* Concurrent diagnosis of interstitial lung disease
* Presence of restrictive pattern on spirometry
* No history of smoking habit
* Individuals not able to provide their written informed consent.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD outpatients with diagnosis of COPD according to the GOLD guidelines (www.goldcopd.org).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of cardiovascular events in COPD patients living with frailty vs non-frail COPD. patients. | 12 and 24 months
  Number of cardiovascular events (including hospital admissions for cardiovascular events) at 12 and 24 months in COPD patients living with frailty vs non-frail COPD patients.

SECONDARY OUTCOMES:
All-cause long-term mortality in COPD patients living with frailty vs non-frail COPD patients. | 12 and 24 months
  All-cause long-term mortality at 12 and 24 months in COPD patients living with frailty vs non-frail COPD patients.
Cardiovascular mortality in COPD patients living with frailty vs non-frail COPD patients. | 12 and 24 months
  Long-term cardiovascular mortality at 12 and 24 months in COPD patients living with frailty vs non-frail COPD patients.
Prevalence of frailty in COPD. | Baseline, at 12 and 24 months
  Prevalence of frailty in COPD.
Deaths due to COPD in COPD patients living with frailty vs non-frail COPD patients. | 12 and 24 months
  Number of deaths due to COPD at 12 and 24 months in COPD patients living with frailty vs non-frail COPD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Alessia Verduri, PhD, Principal Investigator — Respiratory Unit-University of Modena (Italy) - Hospital Policlinico Modena; Alessia Verduri, PhD, Study Director — Respiratory Unit-University of Modena (Italy)-Hospital Policlinico Modena
Locations (1):
- Respiratory Unit - Hospital Policlinico Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Mitnitski AB, Mogilner AJ, Rockwood K. Accumulation of deficits as a proxy measure of aging. ScientificWorldJournal. 2001 Aug 8;1:323-36. doi: 10.1100/tsw.2001.58. PMID 12806071
- [Background] Morley JE, Vellas B, van Kan GA, Anker SD, Bauer JM, Bernabei R, Cesari M, Chumlea WC, Doehner W, Evans J, Fried LP, Guralnik JM, Katz PR, Malmstrom TK, McCarter RJ, Gutierrez Robledo LM, Rockwood K, von Haehling S, Vandewoude MF, Walston J. Frailty consensus: a call to action. J Am Med Dir Assoc. 2013 Jun;14(6):392-7. doi: 10.1016/j.jamda.2013.03.022. PMID 23764209
- [Background] Marengoni A, Vetrano DL, Manes-Gravina E, Bernabei R, Onder G, Palmer K. The Relationship Between COPD and Frailty: A Systematic Review and Meta-Analysis of Observational Studies. Chest. 2018 Jul;154(1):21-40. doi: 10.1016/j.chest.2018.02.014. Epub 2018 Mar 1. PMID 29477493
- [Background] Luo J, Zhang D, Tang W, Dou LY, Sun Y. Impact of Frailty on the Risk of Exacerbations and All-Cause Mortality in Elderly Patients with Stable Chronic Obstructive Pulmonary Disease. Clin Interv Aging. 2021 Apr 13;16:593-601. doi: 10.2147/CIA.S303852. eCollection 2021. PMID 33880018
- [Background] Kennedy CC, Novotny PJ, LeBrasseur NK, Wise RA, Sciurba FC, Benzo RP. Frailty and Clinical Outcomes in Chronic Obstructive Pulmonary Disease. Ann Am Thorac Soc. 2019 Feb;16(2):217-224. doi: 10.1513/AnnalsATS.201803-175OC. PMID 30433830
- [Background] Lee SY, Nyunt MSZ, Gao Q, Gwee X, Chua DQL, Yap KB, Wee SL, Ng TP. Co-occurrence of Physical Frailty and COPD and Association With Disability and Mortality: Singapore Longitudinal Ageing Study. Chest. 2022 May;161(5):1225-1238. doi: 10.1016/j.chest.2021.12.633. Epub 2021 Dec 13. PMID 34914976
- [Background] Galizia G, Cacciatore F, Testa G, Della-Morte D, Mazzella F, Langellotto A, Raucci C, Gargiulo G, Ferrara N, Rengo F, Abete P. Role of clinical frailty on long-term mortality of elderly subjects with and without chronic obstructive pulmonary disease. Aging Clin Exp Res. 2011 Apr;23(2):118-25. doi: 10.1007/BF03351076. PMID 21743290
- [Background] Lahousse L, Ziere G, Verlinden VJ, Zillikens MC, Uitterlinden AG, Rivadeneira F, Tiemeier H, Joos GF, Hofman A, Ikram MA, Franco OH, Brusselle GG, Stricker BH. Risk of Frailty in Elderly With COPD: A Population-Based Study. J Gerontol A Biol Sci Med Sci. 2016 May;71(5):689-95. doi: 10.1093/gerona/glv154. Epub 2015 Sep 9. PMID 26355016
- [Background] Divo M, Cote C, de Torres JP, Casanova C, Marin JM, Pinto-Plata V, Zulueta J, Cabrera C, Zagaceta J, Hunninghake G, Celli B; BODE Collaborative Group. Comorbidities and risk of mortality in patients with chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Jul 15;186(2):155-61. doi: 10.1164/rccm.201201-0034OC. Epub 2012 May 3. PMID 22561964
- [Background] Rockwood K, Song X, MacKnight C, Bergman H, Hogan DB, McDowell I, Mitnitski A. A global clinical measure of fitness and frailty in elderly people. CMAJ. 2005 Aug 30;173(5):489-95. doi: 10.1503/cmaj.050051. PMID 16129869
- [Result] Clegg A, Young J, Iliffe S, Rikkert MO, Rockwood K. Frailty in elderly people. Lancet. 2013 Mar 2;381(9868):752-62. doi: 10.1016/S0140-6736(12)62167-9. Epub 2013 Feb 8. PMID 23395245
- [Derived] Verduri A, Clini E, Carter B, Hewitt J. Influence of frailty on cardiovascular events and mortality in patients with Chronic Obstructive Pulmonary Disease (COPD): Study protocol for a multicentre European observational study. PLoS One. 2024 Jun 25;19(6):e0300945. doi: 10.1371/journal.pone.0300945. eCollection 2024. PMID 38917212
- See also: Global Initiative for Chronic Obstructive Pulmonary Disease (GOLD) — http://www.goldcopd.org